CLINICAL TRIAL: NCT00797888
Title: Bronx A1c: Bring it Down for Health
Acronym: Bronx A1c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: New York City Department of Health and Mental Hygiene (Other Government); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-271; R18DK078077 (NIH)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; behavioral intervention; HbA1c; health disparities
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephonic (Experimental): Tailored telephonic intervention to improve HbA1c for participants in the diabetes registry
  Interventions: Behavioral: telephonic
- Standard registry (Active Comparator): People with diabetes who are in the A1c registry may receive letters from the DOHMH to promote improved A1c and also give lists of bronx resources for healther foof and activites
  Interventions: Behavioral: telephonic

INTERVENTIONS:
Behavioral: telephonic — Between 4-8 phone calls each year for health behavior counseling to improve HbA1c

SUMMARY:
To address and reduce population-attributable risk due to elevated HbA1c, the New York City Department of Health and Mental Hygiene (DOHMH) developed an innovative HbA1c registry, which requires all major laboratories to report HbA1c results electronically. We propose to utilize this registry to conduct a randomized controlled trial addressing the following specific aims: 1) to evaluate the incremental effect of a tiered and tailored, patient-centered telephone intervention, in English and Spanish, on the mean HbA1c levels beyond that achieved with print materials mailed to patients and providers by the DOHMH registry intervention; 2) determine what patient demographic and psychosocial factors mediate the effect of the interventions; and 3) provide estimates of implementation costs of the tiered, tailored telephone intervention for comparison with the print intervention. The study outcome will be change in HbA1c values from the registry records from baseline to one-year post-randomization. A total of 941 individuals with diabetes will be needed to provide 83% power to detect a statistically significant difference (p<0.05) between groups of at least 0.3% in absolute HbA1c. Intervention cost data will be evaluated for translation of findings and scalability. At study end, we will know the extent to which this intervention will improve metabolic control in a low-income, multi-ethnic sample who are part of the DOHMH HbA1c registry in the South Bronx, New York. These findings will inform public health policies and practices in New York City, as well as other urban areas throughout the nation.

DETAILED DESCRIPTION:
Metabolic control of diabetes, measured by hemoglobin A1c (HbA1c), reduces the risk of microvascular complications. Health care providers frequently do not meet standards for managing HbA1c and individuals with diabetes are often not aware of their HbA1c values. To address these issues and reduce population-attributable risk due to elevated HbA1c, the New York City Department of Health and Mental Hygiene (DOHMH) developed an innovative HbA1c registry, which requires all major laboratories to report HbA1c results electronically. We propose to utilize this registry to conduct a randomized controlled trial addressing the following specific aims: 1) to evaluate the incremental effect of a tiered and tailored, patient-centered telephone intervention, in English and Spanish, on the mean HbA1c levels beyond that achieved with print materials mailed to patients and providers by the DOHMH registry intervention; 2) determine what patient demographic and psychosocial factors mediate the effect of the interventions; and 3) provide estimates of implementation costs of the tiered, tailored telephone intervention for comparison with the print intervention. The individual is the unit of sampling, assignment and analysis. After eligibility is assessed and informed consent is obtained by telephone, the individual will be randomly assigned to one of the two groups. The patient telephone intervention will focus on collaborative problem solving for resolving barriers to medication adherence, improving lifestyle behaviors, and communicatiing effectively with their providers. The print materials from the DOHMH will communicate HbA1c results to patients and their providers, with strategies to improve them. The study outcome will be change in HbA1c values from the registry records from baseline to one-year post-randomization. A total of 941 individuals with diabetes will be needed to provide 83% power to detect a statistically significant difference (p<0.05) between groups of at least 0.3% in absolute HbA1c. Psychosocial data on depression, health behaviors, and risk perceptions will be collected by telephone. Intervention cost data will be evaluated for translation of findings and scalability. At study end, we will know the extent to which this intervention will improve metabolic control in a low-income, multi-ethnic sample who are part of the DOHMH HbA1c registry in the South Bronx, New York. These findings will inform public health policies and practices in New York City, as well as other urban areas throughout the nation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be those patients with diabetes who speak English and/or Spanish and reside in the South Bronx.
* Subjects will be adults, > 18 years, with diabetes, who become part of the NYC registry by virtue of having a reported HbA1c >7% to the DOHMH.
* The sampling frame for this study comprises virtually all adults with diabetes in the South Bronx.

Exclusion Criteria:

* Age < 18 years
* A1c < = 7 %
* Refuses informed consent and HIPAA consent
* Cognitive dysfunction as assessed by telephone
* Does not read or speak English or Spanish
* No diabetes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 1 year

SECONDARY OUTCOMES:
diabetes self-care activities | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Gonzalez, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- New York City Department of Health & Mental Hygiene, New York, New York, United States

REFERENCES:
- [Derived] Tabaei BP, Howland RE, Gonzalez JS, Chamany S, Walker EA, Schechter CB, Wu WY. Impact of a Telephonic Intervention to Improve Diabetes Control on Health Care Utilization and Cost for Adults in South Bronx, New York. Diabetes Care. 2020 Apr;43(4):743-750. doi: 10.2337/dc19-0954. Epub 2020 Mar 4. PMID 32132009
- [Derived] Chamany S, Walker EA, Schechter CB, Gonzalez JS, Davis NJ, Ortega FM, Carrasco J, Basch CE, Silver LD. Telephone Intervention to Improve Diabetes Control: A Randomized Trial in the New York City A1c Registry. Am J Prev Med. 2015 Dec;49(6):832-41. doi: 10.1016/j.amepre.2015.04.016. Epub 2015 Jul 29. PMID 26232903
- [Derived] Davis NJ, Schechter CB, Ortega F, Rosen R, Wylie-Rosett J, Walker EA. Dietary patterns in Blacks and Hispanics with diagnosed diabetes in New York City's South Bronx. Am J Clin Nutr. 2013 Apr;97(4):878-85. doi: 10.3945/ajcn.112.051185. Epub 2013 Feb 27. PMID 23446901